CLINICAL TRIAL: NCT00193323
Title: A Randomized Phase III Comparison of Weekly Docetaxel Versus Weekly Docetaxel/Gemcitabine in the Treatment of Elderly or Poor Performance Status Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Weekly Docetaxel Versus Weekly Docetaxel/Gemcitabine in the Treatment of Non-Small Cell Lung Cancer in Elderly Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 52; 104864-450
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2009-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Docetaxel; Gemcitabine

INTERVENTIONS:
Drug: Docetaxel
Drug: Gemcitabine

SUMMARY:
In this randomized trial, we attempt to further define optimal palliative chemotherapy for elderly patients with advanced non-small cell lung cancer by comparing single agent treatment with weekly docetaxel versus combination therapy with weekly docetaxel plus gemcitabine.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will be randomly assigned to one of two treatment arms:

Docetaxel Docetaxel + Gemcitabine

For ever 2 patients treated, 1 will receive treatment A (docetaxel) and 1 will receive treatment B (Docetaxel + Gemcitabine). The study is not blinded so both the patient and the doctor will know which treatment has been assigned.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Biopsy-proven non-small cell lung cancer
* No previous chemotherapy.
* Age > 65 years
* Age < 65 years requires significant assistance to perform activities of daily
* Stage IV disease or stage IIIB disease
* Ability to perform activities of daily living with minimal assistance
* Measurable or evaluable disease
* Adequate bone marrow, liver and kidney
* All patients must sign written informed consent prior to study entry.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Brain metastases
* Meningeal metastases
* Other uncontrolled malignancies
* History of invasive cancer during the last 5 years
* Moderate to severe peripheral neuropathy

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 346
Dates: Start 2001-08; Primary Completion 2006-05 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
median survival
one-year survival.

SECONDARY OUTCOMES:
toxicity

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (1):
- Tennessee Oncology, PLLC, Nashville, Tennessee, United States

REFERENCES:
- [Result] Hainsworth JD, Spigel DR, Farley C, Shipley DL, Bearden JD, Gandhi J, Ann Houston G, Anthony Greco F. Weekly docetaxel versus docetaxel/gemcitabine in the treatment of elderly or poor performance status patients with advanced nonsmall cell lung cancer: a randomized phase 3 trial of the Minnie Pearl Cancer Research Network. Cancer. 2007 Nov 1;110(9):2027-34. doi: 10.1002/cncr.23019. PMID 17823908